CLINICAL TRIAL: NCT00162877
Title: The Role of CYP2C19 Poor Metabolizers and Extensive Metabolizers of PPI in Short-Term Triple Therapy on the Eradication of H. Pylori Infection: Implication of PK/PD Relationships
Brief Title: The Role of CYP2C19 on the Eradication of H. Pylori Infection:Implication of PK/PD Relationships
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 920505; NTUH93S060
Record Dates: First submitted 2005-09-12; First posted 2005-09-13 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2004-01

CONDITIONS: Peptic Ulcer With H. Pylori Infection; Gastritis With H. Pylori Infection
Keywords: rabeprazole, omeprazole, CYP2C19, H. pylori, PK/PD

INTERVENTIONS:
Drug: Rabeprazole vs. Esomeprazole

SUMMARY:
The objective of this trial is to find the rationale and the optimal dose and duration of regimen for the eradication of H. pylori infection using different proton pump inhibitors.

DETAILED DESCRIPTION:
Helicobacter pylori in known to be closely associated with the pathogenesis of gastroduodenal disorders such as peptide ulcer. Eradication of this bacterium is important in the treatment of these diseases as well as in the reduction of the recurrence. The one-week triple therapy with proton pump inhibitors (PPIs) is now considered to be the standard therapies in the treatment of Helicobacter pylori infection, providing more than 80% eradication rates with few adverse effects. PPIs are mainly metabolized by CYP2C19, which is known to exhibit polymorphisms in both its genotype and phenotype. Based on the PK/PD results of our study on PPI, recently, we have proposed that CYP2C19 poor metabolizers might be subject to advantageous conditions, especially after day-4, for the treatment of H. pylori infection when 20 mg rabeprazole was given twice daily. Our results also suggest a possibility to start the triple therapy on day-4 of rabeprazole treatment to ensure the optimal acid suppression effect for antibiotics to exert the bacteriocidal effect. To find the rationale and the optimal dosing regimen for the eradication of H. pylori infection using different proton pump inhibitors, volunteers of four groups would be included in this study. PPI (rabeprazole or esomeprazole) is given for 7 days. Antibiotics are given starting from day-1 or day-4 of PPI dosing. The eradication rate of H. pylori infection and the PK/PD of PPIs are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female dyspeptic patients with H. pylori-positive peptic ulcer or gastritis will be recruited at the university hospital in this study.

Exclusion Criteria:

* 1)Pregnant or lactating female;*2)Patients have endoscopy-based evidence of gastric malignancy, pyloric obstruction, and esophageal stricture requiring dilation, fresh clot, active bleeding, or perforated ulcers;3)Patients requiring anticoagulants or corticosteroid therapy (at dosages greater than the equivalent of prednisone, 10 mg/day);4)Patients with significant impairment of renal function (creatinine>2mg/dl); liver function impairment (AST and ALT 2x upper limit of normal); severe cardiac disease, e.g. angina pectoris, myocardial infarction, cardiac arrhythmia, congestive heart failure (New York Heart Association Functional Classification III and IV) or acute respiratory disease;5)Patients with a history of esophageal and/or gastric varices;6)Use of other investigational drugs within 30 days prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-06; Study Completion 2005-04

PRIMARY OUTCOMES:
the role of CYP2C19 on the eradication of H. pylori infection

SECONDARY OUTCOMES:
implication of PK/PD relationships

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D., Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Department of Internal Medicine, National Taiwan University Hospital, Taipei, Taiwan